CLINICAL TRIAL: NCT00856596
Title: Efficacy Of Sertaconazole 2% (ERTACZO) in the Treatment of Interdigital Tinea Pedis With Once a Day Treatment for 4 Weeks
Brief Title: Once a Day Topical Treatment for Athlete's Foot Fungus Inbetween the Toes in Males and Females
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jamaica Hospital Medical Center (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Jeffrey M. Weinberg, MD, Jamaica Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08023
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Tinea Pedis; Athlete's Foot; Foot Fungus; Ringworm
Keywords: Tinea pedis; Fungus; Pruritus; Dermatophyte; Athlete's foot; Dermatomycosis; Skin manifestation; Infectious skin disease; Foot diseases
MeSH Terms: conditions — Tinea Pedis; Tinea; Pruritus; Dermatomycoses; Skin Manifestations; Skin Diseases, Infectious; Foot Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Males and females with athlete's foot (Other): Male and female subjects with athlete's foot inbetween their toes without nail involvement
  Interventions: Drug: Sertaconazole nitrate cream 2%

INTERVENTIONS:
Drug: Sertaconazole nitrate cream 2% — Once a day topical cream
  Other Names: Ertaczo cream 2%

SUMMARY:
The topical cream, Sertaconazole (Ertaczo), has been FDA approved for the treatment of athlete's foot using twice a day dosing for 4 weeks. This study wants to see if sertaconazole will work equally as well with once a day dosing for 4 weeks for athlete's foot.

DETAILED DESCRIPTION:
The dermatophytes are a group of pathogenic fungi that inhabit and invade keratinized tissue including hair, skin and nails in humans. Infections caused by the three genera of organisms making up the dermatophytes include: Trichophyton, Microsporum and Epidermophyton. Infections due to the dermatophytes are termed dermatophytosis or tinea.

Tinea pedis (athlete's foot) is most commonly caused by Trichophyton rubrum, and less commonly by Trichophyton mentagrophytes and Epidermophyton floccosum.

Tinea infections have been on the rise for variety of reasons including: an aging population, an increase in immunocompromised individuals, increase use of gyms, swimming pools, sports activities, wearing of occlusive footwear, and the organisms themselves becoming more resistant to therapy.

Treatment for tinea pedis usually involves the use of topical therapy with azoles or similar antifungal agents. The efficacy of the topical agent depends on the duration of therapy, type of lesion, the mechanism of action of the drug, and the viscosity, hydrophobicity and acidity of the formulation.

Sertaconazole is a broad spectrum, antifungal agent effective against Candida and dermatophytes. It has also shown antibacterial and anti-inflammatory activity. Skin absorption studies have revealed acceptable therapeutic levels of sertaconazole remained in the skin until 48 hours after application. Half life for drug clearance from the skin is 60 hours. Skin tolerability and phototoxicity studies have revealed sertaconazole to be effective and safe when compared to other topical antifungal agents.

In 2004 sertaconazole nitrate 2% cream, was FDA approved for the topical treatment of interdigital tinea pedis in immunocompetent patients 12 years of age and older, caused by Trichophyton rubrum. Trichophyton mentagrophytes and Epidermophyton floccosum. The approved dosage is twice a day for a total of four weeks to the affected area. This treatment regimen may prove to be difficult for many patients to follow and cause a lower cure rate than would be expected.

It would seem reasonable to postulate that a once a day application would provide adequate therapeutic levels for interdigital tinea pedis based on several previous findings. Acceptable therapeutic levels of drug were maintained in the skin after 48 hours of application and the half-life of the drug is 60 hours. Patient compliance and therefore a higher mycological cure rate and better clinical outcome should theoretically occur with once a day dosing of sertaconazole 2%. Once a day dosing should prevent early discontinuation and better compliance for patients with tinea pedis.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 years of age and over.
2. Women of child bearing age must have a negative urine pregnancy test at Day 0 (baseline) and Day 42 (visit 6) or at the discontinuation visit and must agree to use an acceptable method of contraception during the study.
3. Subjects must have clinical evidence of interdigital tinea pedis of one or both feet characterized by: moderate erythema and scaling and mild pruritis.
4. The clinical diagnosis must be confirmed by a positive KOH preparation, where fungal elements are visible from a skin scraping of the interdigital area of the feet.
5. Fungal cultures obtained at the baseline visit must be positive by day 14 for the subject to remain in the study.
6. All non-study medications not specifically excluded by this protocol may be continued.
7. All chronic diseases must be stable for at least one month.
8. Acute illnesses must be stabilized before enrollment.
9. The subject must be able to understand what is required, read and sign the informed consent, comply with the requirements of this study and adhere to the visit schedule.

Exclusion Criteria:

1. Under 18 years of age.
2. Pregnant or lactating females.
3. Treatment of sertaconazole or an investigational drug within the last 30 days prior to study enrollment.
4. No medications or emollients or foot powders or treatments other than those used in the study are to be applied to the treatment areas.
5. The following medications may not be used during the study:

   * Oral anti-fungals 3 months prior to enrollment
   * Topical anti-fungals to the feet 14 days prior to enrollment
   * Systemic antibiotic or corticosteroid 30 days prior to enrollment
   * Topical corticosteroid 30 days prior to enrollment
   * Use of radiation therapy and/or anti-neoplastic agents within1 year of enrollment
6. Widespread dermatophytosis: moccasin tinea pedis, onychomycosis, oral, vaginal or chronic mucocutaneous candidiasis, bacterial skin infection.
7. Subject who are known or suspected to be immunocompromised.
8. Known sensitivity to any components of the test medication or hypersensitivity to imidazoles.
9. Any disease or condition that may compromise the evaluation of the therapeutic response of tinea pedis to treatment.
10. History of drug or alcohol dependency in the last 6 months.
11. History of atopic or contact dermatitis on the feet.
12. Unstable diabetes mellitus.
13. Subjects who have participated in any previous clinical trial of sertaconazole.
14. Subjects who cannot or will not sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-08 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
To compare the efficacy and safety of sertaconazole 2% cream applied once a day for four weeks in the treatment of patients with KOH positive and culture positive symptomatic interdigital tinea pedis (athlete's foot). | Baseline visit, 1 week, 2 weeks, 4 weeks, 6 weeks

SECONDARY OUTCOMES:
To compare the time to successful clinical and mycological treatment outcomes for sertaconazole 2% cream applied once a day for four weeks in the treatment of patients with KOH positive and culture positive symptomatic interdigital tinea pedis. | Baseline visit, 1 week, 2 weeks, 4 weeks, 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Weinberg, MD, Principal Investigator — Jamaica Hospital Medical Center
Locations (1):
- Jamaica Hospital Medical Center, Jamaica, New York, United States